CLINICAL TRIAL: NCT02525627
Title: A Comparative Study of In-vivo Wear Between 28 mm and 40 mm Metal Heads With Highly Cross Linked (X3) Acetabular Polyethylene Insert in the Hemispherical Trident Cup
Brief Title: A Comparative Study of In-vivo Wear Between 28 mm and 40 mm Metal Heads
Acronym: X3largeheads
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-S-045
Record Dates: First submitted 2015-06-11; First posted 2015-08-17 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trident cup, X3 inserts, 28 mm head (Active Comparator): Equality of 5 year wear in the 28mm and the 40mm metal femoral head sizes. Trident cup in combination with Symax stem or Accolade TMZF stem.
  Interventions: Device: Trident cup, X3 inserts, 28 mm head; Device: Symax stem; Device: Accolade TMZF stem
- Trident cup, X3 inserts, 40 mm head (Active Comparator): Equality of 5 year wear in the 28mm and the 40mm metal femoral head sizes. Trident cup in combination with Symax stem or Accolade TMZF stem.
  Interventions: Device: Trident cup, X3 inserts, 40 mm head; Device: Symax stem; Device: Accolade TMZF stem

INTERVENTIONS:
Device: Trident cup, X3 inserts, 28 mm head — Orthopaedic implant
  Arms: Trident cup, X3 inserts, 28 mm head
Device: Trident cup, X3 inserts, 40 mm head — Orthopaedic implant
  Arms: Trident cup, X3 inserts, 40 mm head
Device: Symax stem — Orthopaedic implant
Device: Accolade TMZF stem — Orthopaedic implant

SUMMARY:
Prospective, single centre, randomized clinical study; series of patients with a 5-years patient evaluation period.

DETAILED DESCRIPTION:
This is a single centre randomized clinical outcomes study. The Symax stem or Accolade TMZF (Titan, Molybdenum, Zirconium, Ferrum) in combination with the Hemispherical Trident cup, X3 inserts, 28 and 40 mm Metal heads are the primary components to be implanted for evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Male and non pregnant female patients between 18-75 years of age.
2. Patients requiring uncemented primary total hip arthroplasty (THA), suitable for the use of the Symax stem
3. Patients with a diagnosis of osteoarthritis (OA), rheumatoid arthritis (RA), avascular necrosis (AVN) or post-traumatic arthritis (TA).
4. Patients who understand the conditions of the study and are willing and able to comply with the post-operative scheduled clinical and radiographic evaluations and the prescribed rehabilitation
5. Patients who signed the specific Informed Consent Form prior to surgery

Exclusion Criteria:

1. Patients who require revision of a previously implanted THA
2. Patients who had a THA on contra-lateral side within the last 1 year.
3. Patients who had a THA on contralateral side more than 1 year ago and the rehabilitation period outcome was considered unsatisfactory or not good. (Patients with contra-lateral THA > 1 year ago with good outcome (Harris Hip Score > 85) can be included in the study).
4. Patients who will need lower limb joint replacement for another joint within one year.
5. Bilaterally operated patient.
6. Patients who have had a prior procedure of acetabular osteotomy.
7. Patients with active or suspected infection.
8. Patients with malignancy - active malignancy
9. Patients with a diagnosed systemic disease that would affect the subject's welfare or overall outcome of the study (i.e. severe osteoporosis, Paget's disease, renal osteodystrophy) or is immunologically suppressed, or receiving steroids in excess of physiologic dose requirements.
10. The patient has a neuromuscular or neurosensory deficit which would limit the ability to assess the performance of the device or the patient has a neurological deficit which interferes with the patient's ability to limit weight bearing or places an extreme load on the implant during the healing period.
11. Female patients planning a pregnancy during the course of the study.
12. Patients with systemic or metabolic disorders leading to progressive bone deterioration.
13. Patients, who as judged by the surgeon, are mentally incompetent or are unlikely to be compliant with the prescribed post-operative routine and follow-up evaluation schedule.
14. Patients with other severe concurrent joint involvements which can affect their outcome.
15. Patients with other concurrent illnesses which are likely to affect their outcome such as sickle cell anaemia, systemic lupus erythematosus, psoriasis, Insulin dependent Type I diabetes or renal disease requiring dialysis.
16. Surgeries to be performed with navigation and/or robot-assisted instruments.
17. Patient with a known sensitivity to device materials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2016-01-12 (Actual); Study Completion 2016-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ide C. Heyligers, MD, Principal Investigator — Atrium Medical Center, Heerlen, The Netherlands
Locations (1):
- Atrium Medical Center, Heerlen, Netherlands

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 40 participants/hips - 6 participants/hips excluded during surgery = 34 participants/hips
Period: Overall Study
Arm/Group | Trident Cup, X3 Inserts, 28 mm Head | Trident Cup, X3 Inserts, 40 mm Head
Started | 16 | 18
Completed | 2 | 5
Not Completed | 14 | 13
Not completed — Revision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Death | 1 | 0
Not completed — Site terminated | 11 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trident Cup, X3 Inserts, 28 mm Head | Trident Cup, X3 Inserts, 40 mm Head | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.67 (4.68) | 62.91 (6.25) | 64.68 (5.87)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data not available for all participants
  Participants
    number analyzed (Participants) | 12 | 13 | 25
    Female | 8 | 10 | 18
    Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  Netherlands | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: To Compare Wear of the Polyethylene X3 Insert Based on Digital Radiographs Using the Hip Analysis Suite (HAS).
Description: Determine equality of 5 year wear in the 28mm and the 40mm metal femoral head sizes using HAS, a software for the determination of polyethylene wear on digital radiographs.
Time Frame: 5 years follow-up
Population: Wear data were not measured at the investigation site.
Arm/Group | Trident Cup, X3 Inserts, 28 mm Head | Trident Cup, X3 Inserts, 40 mm Head
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Harris Hip Score (HHS) Patient Questionnaire
Description: Scores can range from 0 to 100 with 0 being the worst and 100 being the best score. A score of 80-100 is considered good-excellent and a score of less than or equal to 79 is considered fair-poor. 90-100 = excellent 80-89 = good 70-79 = fair 0-69 = poor.
Time Frame: 6 weeks, 3 months, 1, 2 and 5 years
Population: Participants with available data. Overall number of participants analysed is based upon the 6 week population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Trident Cup, X3 Inserts, 28 mm Head | Trident Cup, X3 Inserts, 40 mm Head
Number analyzed (Participants) | 13 | 15
units on a scale
  6 weeks HHS | 82.89 (11.38) | 85.73 (7.91)
  3 months HHS: number analyzed (Participants) | 11 | 14
  3 months HHS | 87.06 (12.03) | 92.60 (4.08)
  1 year HHS: number analyzed (Participants) | 13 | 13
  1 year HHS | 91.71 (6.14) | 92.76 (4.30)
  2 years HHS: number analyzed (Participants) | 10 | 15
  2 years HHS | 90.48 (6.05) | 92.63 (6.81)
  5 years HHS: number analyzed (Participants) | 2 | 5
  5 years HHS | 92.36 (6.56) | 85.95 (21.43)

3. Secondary Outcome: Merle D'Aubergine Score (MdA)
Description: The Merle D'Aubergine-Charnley Score is a simplified clinical scoring system for the hip. The overall score is determined by the sum of scores obtained from each dimension of pain, walking ability and joint mobility. The overall numeric score is given by adding the domain scores. Clinical grades: Excellent, 18, Good 15-17, Fair 13-14, Poor <13.
Time Frame: 6 weeks, 3 months, 1, 2 and 5 years
Population: Merle D'Aubergine Score (MdA) data were not measured at the investigation site.
Arm/Group | Trident Cup, X3 Inserts, 28 mm Head | Trident Cup, X3 Inserts, 40 mm Head
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years post-operative
Arm/Group | Trident Cup, X3 Inserts, 28 mm Head | Trident Cup, X3 Inserts, 40 mm Head
Serious Adverse Events (participants affected / at risk) | 6/16 | 2/18
Other Adverse Events (participants affected / at risk) | 0/16 | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trident Cup, X3 Inserts, 28 mm Head (N=16) | Trident Cup, X3 Inserts, 40 mm Head (N=18)
Luxation of hip prosthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Bladder Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowel Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cardiac Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Intraoperative Trochanter Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Superficial infection (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less